CLINICAL TRIAL: NCT00102934
Title: Treatment Intensification in HIV-1 Patients With Multi-Drug Resistant Virus
Brief Title: Treatment Intensification for HIV Infected Patients With Multi-Drug Resistant Virus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Steven G. Geeks, MD, Department of Medicine, University of California - San Francisco
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5R21AI055273-02 (NIH); Protocol 834; 5R21AI055273-02 (NIH)
Record Dates: First submitted 2005-02-04; First posted 2005-02-07 (Estimated); Last update posted 2008-09-17 (Estimated); Status verified 2008-09

CONDITIONS: HIV Infections
Keywords: HIV; Drug Resistance; Viral Fitness; HIV Specific Immunity; T Cell Activation; Drug Resistant Viremia; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Enfuvirtide

ARMS (1):
- 1 (Experimental): Participants will receive enfuvirtide for 6 months
  Interventions: Drug: Enfuvirtide-intensified HAART

INTERVENTIONS:
Drug: Enfuvirtide-intensified HAART — 90 mg tablet taken orally twice daily
  Other Names: T-20; Fuzeon

SUMMARY:
Drug resistance may develop in HIV infected patients who take anti-HIV drugs, but most patients do well if they continue taking them. The purpose of this study is to test the effectiveness of a short, intensified course of anti-HIV drugs for controlling HIV infection in adults who have virus resistant to multiple drugs.

DETAILED DESCRIPTION:
While an HIV infected patient is taking highly active antiretroviral therapy (HAART), drug-resistant HIV may emerge; however, it has been observed that HIV viral loads while on HAART are usually lower than baseline levels. Expansion of the T cell population during early HAART may explain this phenomenon. It is hoped that a short but aggressive HAART regimen to treatment-experienced patients who have drug-resistant virus will produce immune cells that will better control drug-resistant virus. This study will determine if a 6-month HAART regimen intensified by enfuvirtide (T-20) is effective in eliciting a stronger immune response against drug-resistant virus.

This study will last 48 weeks. All participants will receive T-20 as part of a HAART intensification regimen; HAART other than T-20 will not be provided by the study. There will be 17 study visits. Prior to beginning treatment intensification, participants will have weekly study visits for three weeks. Once treatment intensification has started, participants will be followed weekly for four weeks, then weekly for four weeks after treatment intensification, then monthly thereafter. Blood collection will occur at each visit.

ELIGIBILITY:
Inclusion Criteria:

* HIV viral load of more than 1000 copies/ml
* On stable antiretroviral therapy
* Have multidrug resistance

Exclusion Criteria:

* Require immunomodulatory drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-03; Primary Completion 2005-12 (Actual); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
HIV viral load | Throughout study

SECONDARY OUTCOMES:
Frequency of HIV-specific T cells | Thoughout study

CONTACTS AND LOCATIONS:
Overall Officials: Steven G. Deeks, MD, Principal Investigator — Department of Medicine, University of California - San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States